CLINICAL TRIAL: NCT04767802
Title: A Phase 2 Study of the Hepcidin Mimetic PTG-300 in Patients With Polycythemia Vera and Elevated Hematocrit (PACIFIC)
Brief Title: PTG-300 in Patients With Polycythemia Vera and Elevated Hematocrit
Acronym: PACIFIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTG-300-08
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Polycythemia Vera
Keywords: PV
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PTG-300 (Experimental): Evaluate PTG-300's efficacy and safety in subjects with PV and baseline elevated hematocrit.
  Interventions: Drug: PTG-300

INTERVENTIONS:
Drug: PTG-300 — Hepcidin mimetic
  Other Names: Rusfertide

SUMMARY:
This is an open label, single arm trial of PTG-300 in subjects with PV who are newly diagnosed or for whom current therapy is not sufficient to control their hematocrit and have hematocrit >48% prior to dosing. The PTG-300 dose and schedule may be adjusted every 2 to 4 weeks to maintain hematocrit <45% with a target of <43%. Subjects may receive PTG-300 treatment for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Known diagnosis of polycythemia vera.
2. Hematocrit >48% before dosing.
3. Evidence of hematocrit >48% three or more times in the 28 weeks before dosing or five or more times in 52 weeks before dosing (except for newly diagnosed patients).
4. Clinically reasonable alternative causes for erythrocytosis have been evaluated and excluded.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.

Exclusion Criteria:

1. Clinically significant thrombosis (e.g., deep vein thrombosis or splenic vein thrombosis) within 3 months of Screening.
2. Active or chronic bleeding within 4 weeks of Screening.
3. Meets the criteria for post-PV myelofibrosis as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT).
4. Infection requiring hospitalization or intravenous antimicrobial therapy, or opportunistic infection within 3 months of dosing; any infection requiring systemic antimicrobial therapy within 4 weeks of dosing. Prophylactic antibiotics are allowed.
5. Any serious or unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the subject from properly providing informed consent or any condition which would jeopardize compliance with the study.
6. Known primary or secondary immunodeficiency.
7. Known positive for active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
8. Any surgical procedure requiring general anesthesia within 1 month prior to Screening or planned elective surgery during the study.
9. History of invasive malignancies within the last 2 years, except non-melanoma skin cancer and localized curatively treated prostate cancer or cervical cancer.
10. Current or recent history of alcohol dependence or illicit drug use within 1 year prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluate PTG-300's efficacy in subjects with PV and baseline elevated hematocrit. | Estimate the proportion of subject with a hematocrit less than 45% at Week 16
  Proportion of subjects with hematocrit <45%

SECONDARY OUTCOMES:
Safety of PTG-300 | Week 52
  Proportion of Subjects Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (8):
- Malaysia (5):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Raja Perempuan Zainab, Kota Bharu, Kelantan
  - Hospital Raja Permaisuki Bainun, Ipoh, Perak
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Ampang, Ampang, Selangor
- South Korea (3):
  - Gachon University Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Catholic University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No